CLINICAL TRIAL: NCT06526273
Title: The PILI 'Āina Project
Brief Title: PILI 'Āina Household
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILI 'Āina 2; R01HL168858 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-07-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Hypertension; Dyslipidemias; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PILI 'Āina (Experimental): Participants will receive the 3-month adapted Diabetes Prevention Program's Lifestyle Intervention. At 3 months, participants randomized to the PILI 'Āina intervention will receive a 6-month intervention centered around the use of a raised-bed home garden as the means of engaging household members to 1) increase their access to and intake of vegetables, 2) learn culturally relevant ways of preparing/cooking fresh vegetables through hands-on cooking lessons with local experts, and 3) build family cohesion through family bonding activities. The participating households will be given all the equipment and materials (e.g., soil, seeds, instructions, setup of equipment) needed to grow their vegetables using their raised-bed home garden box throughout the entire study. The investigators will provide seeds for the vegetables that can grow in a relatively short period (i.e., within 6 weeks). All lessons will be delivered by a trained community health worker .
  Interventions: Behavioral: PILI 'Āina
- Control (Active Comparator): Participants randomized to the control group will receive monthly untailored health education information and links to community resources from the community health worker via United States Postal Service or electronic messaging. Examples include information on food assistance programs, farmers markets, cultural events, and physical activity events.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: PILI 'Āina — Participants will receive the 3-month adapted Diabetes Prevention Program's Lifestyle Intervention. These lessons will be delivered by a trained community health worker. At 3 months, participants randomized to the PILI 'Āina intervention will receive a 6-month intervention centered around the use of a raised-bed home garden as the means of engaging household members to 1) increase their access to and intake of vegetables, 2) learn culturally relevant ways of preparing/cooking fresh vegetables through hands-on cooking lessons with local experts, and 3) build family cohesion through family bonding activities. Participants will be given all the equipment and materials (e.g., soil, seeds, instructions, setup of equipment) needed to grow their vegetables using their raised-bed home garden box throughout the entire study. They will receive seeds for the vegetables that can grow in a relatively short period (i.e., within 6 weeks).
  Arms: PILI 'Āina
Other: Control — Participants will receive the 3-month adapted Diabetes Prevention Program's Lifestyle Intervention. These lessons will be delivered by a trained community health worker based on previously tested materials and protocols. At 3 months, participants randomized to the control group will receive monthly untailored health education information and links to community resources from the community health worker via United States Postal Service or electronic messaging. Examples include information on food assistance programs, farmers' markets, cultural events, and physical activity events.
  Arms: Control

SUMMARY:
Native Hawaiians' traditional lifestyles and diets ensured the mutual health and well-being of the land and its inhabitants, which stand in stark contrast to the disproportionately high prevalence of diet-related, cardiometabolic diseases they experience today. In this project, the investigators will adapt and test an evidence-based multilevel intervention entitled PILI 'Āina to improve the self-management of prevalent cardiometabolic diseases and reduce risk factors for developing new diet-related illnesses and implement and evaluate the impact and sustainability of community-wide cooking demonstrations. The objectives of this project are to optimize the effectiveness and sustainability of PILI 'Āina, improve diet quality, cardiometabolic markers, promote traditional Native Hawaiian diets, and improve social cohesion.

DETAILED DESCRIPTION:
The investigators will conduct a group-randomized controlled trial to test the effectiveness of PILI Aina for improving diet and health at the individual and household levels compared to a Diabetes Prevention Program Lifestyle Intervention only group. The investigators will enroll 180 Native Hawaiian adults with overweight or obesity and at least 1 other diet-related cardiometabolic condition (Type 2 diabetes, pre-diabetes, hypertension, pre-hypertension, dyslipidemia). These index participants will receive the 3-month educational program and then be randomized at the household level to the 6-month PILI Aina intervention or to a control group. Data collection will occur at baseline and 3, 9, and 12 months. Other adult household members will be invited to participate in data collection at the same time to evaluate household-level effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (looking for older adults)
* Native Hawaiian resident in a participating homestead
* Overweight or obese (BMI ≥ 25 kg/m^2)
* Prior diagnosis of T2D or pre-diabetes, hypertension, and/or dyslipidemia (LDL cholesterol ≥ 130 mg/dL)
* Capable of 150 minutes of moderate physical activity (e.g., brisk walking) per week
* Willing and able to participate in all aspects of the individual and household-level intervention
* Fluent in written and spoken English

Exclusion Criteria:

* No children
* Pregnancy
* Serious illness such as cancer or chronic pain that may contraindicate full participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Diet Quality | Baseline, 3 month, 9 month, 12 month
  To measure diet quality, research staff will collect participants' 24-hour dietary recall by using the Modified 3-Pass Method. They will record diet information, and analysis will be performed by the Pacific Tracker (PacTrac) Program, 4th edition, developed at the University of Hawaii Cancer Center to analyze diets common in Hawai'i. It generates a "healthy eating index" (from 0 = least healthy to 100 = healthiest) shown to have good validity and reliability. Continuous values of the overall score will constitute our primary outcome, but the investigators will also evaluate scores for subscales (diet adequacy, moderation). The investigators will also assess diet quality and patterns by comparing servings consumed for each food group (vegetables, fruits, grains, dairy, and protein) to the United States Department of Agriculture (USDA) dietary guidelines.
Weight | Baseline, 3 month, 9 month, 12 month
  The investigators will measure weight (with clothing but without shoes) to the nearest 0.1 kilograms on an electric digital scale (Tanita model BSB800AS, Tokyo, Japan). Scales will be calibrated monthly.
Height | Baseline, 3 month, 9 month, 12 month
  The investigators will use a portable stadiometer (SECA Road Rod) to record the average of 2 measurements of height to the nearest 0.1 cm. Scales will be calibrated monthly.
Blood pressure | Baseline, 3 month, 9 month, 12 month
  Blood pressure will be collected with a mercury sphygmomanometer or with a portable automatic blood pressure device (Omron©HEM-907XL, Omron Healthcare) previously used with Native Hawaiians (NHs) to capture changes in blood pressure over time reliably. For both methods, study staff will be trained and certified with standard protocols that involve taking 3 measurements and using the last 2 to obtain each participant's average systolic and diastolic blood pressure (mm Hg). Systolic and diastolic blood pressure will be measured as continuous mm Hg and binary hypertension indicators (≥ 130 systolic or ≥ 80 mm Hg diastolic).
hemoglobin A1c | Baseline, 3 month, 9 month, 12 month
  Hemoglobin A1c will be measured by DCA Vantage portable analyzers, using blood samples by fingerstick. Results are available in 5 minutes and will be returned to participants. A1c values will be recorded both as a continuous value (%) to the tenths digit and as a binary indicator of A1c < 8%.
Lipids | Baseline, 3 month, 9 month, 12 month
  Lipids will be measured by Alere Cholestech LDX portable analyzers, using blood samples by fingerstick. Results are available in 5 minutes and will be returned to participants. Lipids (Low-Density Lipoproteins [LDL] and High-Density Lipoproteins [HDL]) will be measured as continuous mg/dL and as binary indicators of healthy cholesterol levels (LDL ≤ 130; HDL ≥ 40).

SECONDARY OUTCOMES:
Food Insecurity | Baseline, 3 month, 9 month, 12 month
  Food insecurity will be measured by the 10-item Household Food Security Survey Module, which captures the qualitative and quantitative dimensions of household food supply, including psychological and behavioral responses of household members, and generates a binary indicator of food insecurity at the household level. The responses and scores range from 1-often true, 2-sometimes true, 3-never true. Higher scores indicate low food insecurity.
Food literacy | Baseline, 3 month, 9 month, 12 month
  Food literacy, defined as the ability to make healthy food choices in different settings and situations, will be assessed by the 11-item self-perceived food literacy scale, which encompasses knowledge, skills, and behaviors pertinent to planning, selecting, preparing, and eating healthy food. The responses and scores range from 1-not at all/never, 2-disagree, 3-slightly disagree, 4- slightly agree, 5-yes/always. Higher scores indicate greater food literacy.
Nutrition Environment | Baseline, 3 month, 9 month, 12 month
  The perceived 9-item nutrition environment will be measured by the Gustafson Perceived Nutrition Environment Measures questionnaire, which examines perceived access and availability of healthy foods within ~1 mile of the participant's home, and the availability and affordability of produce in the participant's primary food store. The responses and scores vary depending on the question including 0- disagree, 1-agree, and 0-not important, 1-slightly important, 2-moderately important, 3- important, 4-very important. Higher scores indicate higher perceived access and availability of food.
Household food patterns | Baseline, 3 month, 9 month, 12 month
  Household food patterns will be measured by 4 questions that assess the frequency of meal planning, eating meals with household members, bringing prepared restaurant foods home, and preparing meals with household members. The responses and scores range from 1- 1 day, 2- 2-3 days, 3- 4-5 days, 4- 6 days, 5- 7 days. Higher scores indicate greater household food patterns.
Social support | Baseline, 3 month, 9 month, 12 month
  Social support for a healthy diet will be measured as the perceived support that people who make dietary changes receive from family and friends. An 11-item questionnaire on social support will be used to ask participants' perceived level of support from friends and family regarding diet choices. The responses and scores range from 1-strongly disagree, 2-somewhat disagree, 3-neutral, 4-somewhat agree, and 5-strongly agree. Higher scores indicate greater social support.
Medications | Baseline, 3 month, 9 month, 12 month
  Name and dosage for prescription medications for type 2 diabetes, hypertension, dyslipidemia, or cardiovascular disease will be recorded from containers brought to data collection visits.
Physical Activity | Baseline, 3 month, 9 month, 12 month
  The 3-item Physical Activity Questionnaire, which has been used with Native Hawaiians, will assess exercise frequency during the past month. It contains 3 items that assess moderate and vigorous exercise and changes in activity levels. The responses and scores vary depending on the question, including 0- rarely or never, 1- 2-3 times over the month, 2- about once a week, 3- 2-4 times a week, 4- more than 4 times a week. Higher scores indicate greater physical activity.
Diet self-efficacy | Baseline, 3 month, 9 month, 12 month
  The 11-item Diet Self Efficacy Scale will measure self-efficacy in avoiding tempting high caloric food and managing social and internal cues and negative emotions. The responses and scores range from 1-strongly disagree, 2-somewhat disagree, 3-neutral, 4-somewhat agree, and 5-strongly agree. Higher scores indicate greater self-efficacy with diet.

OTHER OUTCOMES:
Demographic Data- Date of Birth | Baseline
  Date of birth:
  * Month
  * Day
  * Year
Demographic Data- Biological Sex | Baseline
  Biological Sex:
  * Female
  * Male
Demographic Data- Marital status | Baseline
  Marital Status:
  * Never married
  * Currently married
  * Divorced or separated
  * Widow/widower
  * Domestic partnership/other
Demographic Data- Employment | Baseline
  Employment:
  * Full time
  * Part-time
  * Unemployed
  * Self-employed
  * Retired
  * Unable to work/other
  * Household caretaker
Demographic Data- Education | Baseline
  Education:
  * Less than high school
  * High school diploma/General Education Diploma (GED)
  * Some college/technical training
  * College degree
  * Graduate/professional degree
Demographic Data- Ethnic ancestry | Baseline
  Ethnic Ancestry:
  * Caucasian
  * Chinese
  * Filipino
  * Hawaiian
  * Latino
  * Japanese
  * Korean
  * Marshallese
  * Micronesian (specify)
  * Native American
  * Portuguese
  * Samoan
  * Other (specify)
Demographic Data- Household income | Baseline
  Household Income:
  * Under $49,999
  * $50,000-$74,999
  * $75,000-$99,999
  * $100,000-$124,999
  * Over $125,000
  Household income will be classified according to the US Census Bureau's poverty threshold by using a dichotomous variable. Participation in public assistance programs (e.g., Temporary Assistance for Needy Families, Supplemental Nutrition Assistance Program) will also be recorded.
Demographic Data- Household Composition | Baseline
  Household Composition:
  1. Who lives in the participants house full-time? (50% or more time spent in-house)
  * Parents
  * Children
  * Grandparents/great-grandparents
  * Other family members
    a. Of those people, what are their ages and genders?
  * Male: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
  * Female: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
  * Number of other/non-binary: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
Smoking/alcohol | Baseline, 3 month, 9 month, 12 month
  Tobacco and alcohol use will be measured by using a measure developed by Dr. Kaholokula for PILI 'Ohana.
Cultural identity | Baseline, 3 month, 9 month, 12 month
  Cultural factors will be measured by the 4-item Cultural Identity Scale that will assess the degree of identification with NH cultural heritage. The responses and scores range from 0-not at all knowledgeable, 1- somewhat not knowledgeable, 2-neutral or no response, 3-somewhat knowledgeable, and 4-very knowledgeable. Higher scores indicate greater cultural identity.
Neighborhood environment | Baseline, 3 month, 9 month, 12 month
  Neighborhood environment will be measured by the 17-item modified Neighborhood Level Stressors Scale, which assesses participants' perceptions of 4 neighborhood dimensions (i.e., walkability, availability of healthy food, safety, and social cohesion). The responses and scores range from 1-strongly disagree, 2-somewhat disagree, 3- neutral, 4-somewhat agree, 5-strongly agree. Higher scores indicate low neighborhood level stressors.
Comorbidities | Baseline, 3 month, 9 month, 12 month
  Existing comorbidities will be measured as whether the participant has ever been told by a healthcare professional that they have had a heart attack, heart failure, stroke, or chronic kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Ing, DrPH, Principal Investigator — University of Hawaii
Locations (2):
- United States (2):
  - Kula no nā Po'e Hawai'i, Honolulu, Hawaii
  - Kapolei Community Development Corporation, Kapolei, Hawaii

IPD SHARING:
Plan to Share IPD: No